CLINICAL TRIAL: NCT03029819
Title: iQuit Mindfully: A Randomized Controlled Trial of Mindfulness-based Smoking Cessation Enhanced With Mobile Technology
Brief Title: iQuit Mindfully: Text Messaging for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Utah (Other); The Catholic University of America (Other); George Washington University (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Claire Spears, Assistant Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23AT008442 (NIH); K23AT008442 (NIH)
Record Dates: First submitted 2017-01-16; First posted 2017-01-24 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Addiction Treatment (MBAT) (Active Comparator): Nicotine patch; self-help guide; MBAT
  Interventions: Behavioral: Mindfulness-based Addiction Treatment; Behavioral: Self-Help guide; Drug: Nicotine Patch
- iQuit Mindfully (Experimental): Nicotine patch; self-help guide; MBAT; text messaging
  Interventions: Behavioral: Mindfulness-based Addiction Treatment; Behavioral: iQuit Mindfully; Behavioral: Self-Help guide; Drug: Nicotine Patch

INTERVENTIONS:
Behavioral: Mindfulness-based Addiction Treatment — Mindfulness-based Addiction Treatment (MBAT) consists of 8 weekly 2-hour sessions that teach mindfulness and cognitive-behavioral strategies for smoking cessation (Wetter et al., 2009).
Behavioral: iQuit Mindfully — iQuit Mindfully involves text messages on each day between treatment sessions. The text messages provide mindfulness and cognitive-behavioral strategies and support for smoking cessation.
  Other Names: Mindfulness-based text messaging for smoking cessation
  Arms: iQuit Mindfully
Behavioral: Self-Help guide — Self-help materials for smoking cessation are based on the Treating Tobacco Use and Dependence Clinical Practice Guideline (Fiore et al. Clinical practice guideline for treating tobacco use and dependence, 2008).
Drug: Nicotine Patch — Patch therapy (beginning the week before quit day) for participants who smoke >10 cigarettes/day will consist of 4 weeks of 21 mg patches, 1 week of 14 mg patches, and 1 week of 7 mg patches. Patch therapy for participants who smoke 5-10 cigarettes/day will consist of 4 weeks of 14 mg patches and 2 weeks of 7 mg patches.
  Other Names: Generic Nicotine Patch

SUMMARY:
The purpose of this study is to investigate text messaging as a way to enhance mindfulness-based treatment for smoking cessation.

DETAILED DESCRIPTION:
This study is a pilot investigation of mindfulness-based smoking cessation treatment incorporating between-session text messaging ("iQuit Mindfully"). Participants will be randomly assigned to one of two groups: Mindfulness-based Addiction Treatment (MBAT) or iQuit Mindfully (MBAT with the addition of between-session text messages).

All participants will receive in-person group treatment based on the 8-week MBAT protocol in addition to nicotine patch therapy and self-help materials. Participants assigned to iQuit Mindfully will receive additional support via text messaging. Assessments will occur at baseline, at each of the weekly in-person visits, at end of treatment, and at 1-month follow-up. Feasibility, smoking abstinence, mindfulness practice, and indicators of tobacco dependence and psychological well-being will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* current smoker with history of >5 cigarettes/day for past year (and expired carbon monoxide >6 parts per million [ppm])
* motivated to quit within next 30 days
* valid home address in the greater Atlanta, Georgia area
* functioning telephone number
* own a mobile phone with text messaging capacity
* can speak, read, and write in English
* at least a sixth-grade level of health literacy

Exclusion Criteria:

* contraindication for nicotine patch
* active substance abuse/dependence
* regular use of tobacco products other than cigarettes
* current use of tobacco cessation medications
* pregnancy or lactation
* household member enrolled in the study
* current diagnosis of schizophrenia or bipolar disorder, or use of antipsychotic medications
* clinically significant depressive symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire A Spears, Ph.D., Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

REFERENCES:
- [Background] Vidrine JI, Spears CA, Heppner WL, Reitzel LR, Marcus MT, Cinciripini PM, Waters AJ, Li Y, Nguyen NT, Cao Y, Tindle HA, Fine M, Safranek LV, Wetter DW. Efficacy of mindfulness-based addiction treatment (MBAT) for smoking cessation and lapse recovery: A randomized clinical trial. J Consult Clin Psychol. 2016 Sep;84(9):824-838. doi: 10.1037/ccp0000117. PMID 27213492
- [Background] Clinical Practice Guideline Treating Tobacco Use and Dependence 2008 Update Panel, Liaisons, and Staff. A clinical practice guideline for treating tobacco use and dependence: 2008 update. A U.S. Public Health Service report. Am J Prev Med. 2008 Aug;35(2):158-76. doi: 10.1016/j.amepre.2008.04.009. PMID 18617085
- [Derived] Spears CA, Abroms LC, Glass CR, Hedeker D, Eriksen MP, Cottrell-Daniels C, Tran BQ, Wetter DW. Mindfulness-Based Smoking Cessation Enhanced With Mobile Technology (iQuit Mindfully): Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jun 24;7(6):e13059. doi: 10.2196/13059. PMID 31237242

RESULTS

PARTICIPANT FLOW:
Groups:
- Mindfulness-based Addiction Treatment (MBAT): Nicotine patch; self-help guide; MBAT
  Mindfulness-based Addiction Treatment: Mindfulness-based Addiction Treatment (MBAT) consists of 8 weekly 2-hour sessions that teach mindfulness and cognitive-behavioral strategies for smoking cessation (Wetter et al., 2009).
  Self-Help guide: Self-help materials for smoking cessation are based on the Treating Tobacco Use and Dependence Clinical Practice Guideline (Fiore et al., 2008).
  Nicotine Patch: Patch therapy (beginning the week before quit day) for participants who smoke >10 cigarettes/day will consist of 4 weeks of 21 mg patches, 1 week of 14 mg patches, and 1 week of 7 mg patches. Patch therapy for participants who smoke 5-10 cigarettes/day will consist of 4 weeks of 14 mg patches and 2 weeks of 7 mg patches.
- iQuit Mindfully: Nicotine patch; self-help guide; MBAT; text messaging
  Mindfulness-based Addiction Treatment: Mindfulness-based Addiction Treatment (MBAT) consists of 8 weekly 2-hour sessions that teach mindfulness and cognitive-behavioral strategies for smoking cessation (Wetter et al., 2009).
  iQuit Mindfully: iQuit Mindfully involves text messages on each day between treatment sessions. The text messages provide mindfulness and cognitive-behavioral strategies and support for smoking cessation.
  Self-Help guide: Self-help materials for smoking cessation are based on the Treating Tobacco Use and Dependence Clinical Practice Guideline (Fiore et al., 2008).
  Nicotine Patch: Patch therapy (beginning the week before quit day) for participants who smoke >10 cigarettes/day will consist of 4 weeks of 21 mg patches, 1 week of 14 mg patches, and 1 week of 7 mg patches. Patch therapy for participants who smoke 5-10 cigarettes/day will consist of 4 weeks of 14 mg patches and 2 weeks of 7 mg patches.
Period: Overall Study
Arm/Group | Mindfulness-based Addiction Treatment (MBAT) | iQuit Mindfully
Started | 33 | 39
Completed | 30 | 33
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 3 | 5
Not completed — Removed due to disruptive behavior | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 72 participants were enrolled in the study. However, one participant was removed due to disruptive behavior in the in-person group treatment, for a final analytic sample of 71 (33 in MBAT and 38 in iQuit Mindfully).
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-based Addiction Treatment (MBAT) | iQuit Mindfully | Total
Number analyzed (Participants) | 33 | 38 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.6 (12.0) | 45.6 (12.4) | 45.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 13 | 21 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 31 | 37 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 34 | 50
  White | 11 | 4 | 15
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 1 | 0 | 1
Baseline cigarettes per day [Mean (Standard Deviation); unit: Cigarettes per day] | 18.8 (9.3) | 14.4 (9.4) | 16.5 (9.6)

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence
Description: Number of participants who abstained from smoking (based on self-reported 7-day abstinence, which is biochemically verified by expired carbon monoxide <6 parts per million (ppm)
Time Frame: End of Treatment (8 weeks)
Population: Available data for smoking abstinence were analyzed because coding missing data as smoking can severely bias results. Accordingly, the overall number of participants analyzed for smoking abstinence was 55.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-based Addiction Treatment (MBAT) | iQuit Mindfully
Number analyzed (Participants) | 24 | 31
Participants | 4 | 8
Statistical Analysis 1: Comparison: Mindfulness-based Addiction Treatment (MBAT) vs iQuit Mindfully; Test type: Superiority; p = .52, Chi-squared

2. Secondary Outcome: Participant Engagement
Description: Number of participants who respond to interactive text messages
Time Frame: Over the 8-week treatment period
Population: Only participants in the iQuit Mindfully condition were included in this analysis because MBAT participants did not receive text messages.
Measure: Count of Participants; unit: Participants
Groups:
- iQuit Mindfully: Nicotine patch; self-help guide; MBAT; text messaging
  Mindfulness-based Addiction Treatment (MBAT) consists of 8 weekly 2-hour sessions that teach mindfulness and cognitive-behavioral strategies for smoking cessation.
  iQuit Mindfully: iQuit Mindfully involves text messages on each day between treatment sessions. The text messages provide mindfulness and cognitive-behavioral strategies and support for smoking cessation.
  Self-Help guide: Self-help materials for smoking cessation are based on the Treating Tobacco Use and Dependence Clinical Practice Guideline.
  Nicotine Patch: Patch therapy (beginning the week before quit day) for participants who smoke >10 cigarettes/day will consist of 4 weeks of 21 mg patches, 1 week of 14 mg patches, and 1 week of 7 mg patches. Patch therapy for participants who smoke 5-10 cigarettes/day will consist of 4 weeks of 14 mg patches and 2 weeks of 7 mg patches.
Arm/Group | Mindfulness-based Addiction Treatment (MBAT) | iQuit Mindfully
Number analyzed (Participants) | 0 | 38
Participants |  | 34

3. Secondary Outcome: Participant Ratings
Description: Perceived Text Message Helpfulness (minimum value 1 ["not at all helpful"], maximum value 10 ["extremely helpful"], higher scores mean better outcome)
Time Frame: End of Treatment (8 weeks)
Population: Only participants in the iQuit Mindfully condition were included in this analysis because those in MBAT did not receive text messages.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- iQuit Mindfully: Nicotine patch; self-help guide; MBAT; text messaging
  Mindfulness-based Addiction Treatment: Mindfulness-based Addiction Treatment (MBAT) consists of 8 weekly 2-hour sessions that teach mindfulness and cognitive-behavioral strategies for smoking cessation.
  iQuit Mindfully: iQuit Mindfully involves text messages on each day between treatment sessions. The text messages provide mindfulness and cognitive-behavioral strategies and support for smoking cessation.
  Self-Help guide: Self-help materials for smoking cessation are based on the Treating Tobacco Use and Dependence Clinical Practice Guideline.
  Nicotine Patch: Patch therapy (beginning the week before quit day) for participants who smoke >10 cigarettes/day will consist of 4 weeks of 21 mg patches, 1 week of 14 mg patches, and 1 week of 7 mg patches. Patch therapy for participants who smoke 5-10 cigarettes/day will consist of 4 weeks of 14 mg patches and 2 weeks of 7 mg patches.
Arm/Group | Mindfulness-based Addiction Treatment (MBAT) | iQuit Mindfully
Number analyzed (Participants) | 0 | 38
units on a scale |  | 8.0 (2.4)

4. Secondary Outcome: Attrition
Description: Number of participants who do not attend end-of-treatment session
Time Frame: End of treatment (8 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-based Addiction Treatment (MBAT) | iQuit Mindfully
Number analyzed (Participants) | 33 | 38
Participants | 9 | 8

5. Other Pre Specified Outcome: Number of Cigarettes Smoked Per Day
Description: Self-reported number of cigarettes smoked per day (questionnaire)
Time Frame: End of treatment (8 weeks)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Weekly Mindfulness Practice
Description: Self-reported average weekly mindfulness practice (questionnaire)
Time Frame: Throughout treatment period (8 weeks)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Self-reported Mindfulness and Psychological Functioning
Description: Mindfulness, affect, self-efficacy, dependence, and withdrawal symptoms (questionnaire)
Time Frame: End of treatment (8 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Reported over the period of treatment (8 weeks) and 1 month follow-up, for a total of 12 weeks.
Arm/Group | Mindfulness-based Addiction Treatment (MBAT) | iQuit Mindfully
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/39
Other Adverse Events (participants affected / at risk) | 7/33 | 5/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mindfulness-based Addiction Treatment (MBAT) (N=33) | iQuit Mindfully (N=39)
Mild nicotine patch side effects (General disorders) | 7 | 5 — Mild nicotine patch side effects (itching, nausea, abnormal dreams, nervousness)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03029819/Prot_SAP_000.pdf